CLINICAL TRIAL: NCT00487500
Title: Affective and Cognitive Consequences of ECT
Brief Title: Comparing the Effects of Four Types of Electroconvulsive Therapy on Mood and Thinking in People With Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: #3482; 5R01MH035636 (NIH)
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2007-06

CONDITIONS: Depression
Keywords: Major Depressive Disorder; Electroconvulsive Therapy
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ultrabrief, Right Unilateral ECT (Experimental): Right unilateral ECT administered with an ultrabrief pulse width (0.3 ms), at a dose 6 times the initial seizure threshold
  Interventions: Device: Electroconvulsive Therapy (ECT)
- Ultrabrief, Bilateral ECT (2.5 X ST) (Experimental): Bilateral (frontotemporal) ECT with an ultrabrief pulse width with dosage 2.5 times the initial seizure threshold
  Interventions: Device: Electroconvulsive Therapy (ECT)
- Brief Pulse, Right Unilateral ECT (Active Comparator): Right unilateral ECT, with a standard brief pulse (1.5 ms), with dosage 6 times the initial seizure threshold
  Interventions: Device: Electroconvulsive Therapy (ECT)
- Brief Pulse, Bilateral ECT (Active Comparator): Bilateral (frontotemporal) ECT with a standard brief pulse (1.5 ms), with dosage 2.5 times the initial seizure threshold
  Interventions: Device: Electroconvulsive Therapy (ECT)

INTERVENTIONS:
Device: Electroconvulsive Therapy (ECT) — Electroconvulsive therapy involves applying a small electrical charge to the scalp while the patient is anesthetized and provoking a short-lasting generalized seizure
  Other Names: shock therapy

SUMMARY:
This study will compare four types of electroconvulsive therapy to determine if they differ in their effects on mood, thinking, brain activity, and biochemistry in people with major depressive disorder.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a serious condition that can interfere with a person's ability to work, study, sleep, eat, and enjoy activities that were once pleasurable. Depression may occur only once in a lifetime, but usually occurs several times. There are several types of medications and therapies that have been successful in improving symptoms of depression. Electroconvulsive therapy (ECT) has been particularly successful in treating individuals whose depression is severe or life threatening or who cannot take antidepressant medication. In ECT, electrodes are placed at precise locations on the head to deliver electrical impulses. The stimulation causes a brief seizure within the brain. The person receiving ECT does not consciously experience the electrical stimulus and does not feel pain. This study will compare four types of ECT to determine if they differ in their effects on mood, thinking, brain activity, and biochemistry in people with MDD.

Participants in this double-blind study will be randomly assigned to receive one of four types of ECT. Treatments will occur three times a week for 2 to 6 weeks, depending on each participant's individual needs. All participants will stop taking any psychiatric medications at least 5 days before receiving ECT. Before beginning each ECT session, participants will be interviewed by study staff about their current psychiatric condition, any psychological problems they have had, any history of psychological problems in their families, their medical history, and their attitudes about receiving ECT. A family member may also be asked to participate in some interviews. In addition, before each treatment, monitoring sensors will be placed on each participant's head and other areas of the body and a blood pressure cuff will be placed on an arm. These devices will be used to monitor each participant's brain waves, heart, and blood pressure before, during, and after treatment.

Because ECT entails the use of general anesthesia, participants will not eat for at least 8 hours before each treatment. An intravenous catheter will be placed in participants' arms to administer the anesthesia and a muscle relaxant. Just before receiving ECT, participants will be asked to remember a set of information. Upon waking after treatment, participants will be asked to recall or recognize this material and complete a set of brief neuropsychological tasks. Electroencephalogram (EEG) tests (to measure electrical activity of the brain), transcranial magnetic stimulation (TMS) (to measure muscle activity), blood collection, and magnetic resonance imaging (MRI) tests (to image the inside of the body) will be performed at selected sessions and follow-up visits to assess outcomes. Follow-up interviews will be held via telephone every 2 weeks for 2 months post-treatment, and then monthly for the remainder of the year. Follow-up neuropsychological tests will also be administered at Months 2, 4, and 6 post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder
* Pretreatment score of at least 18 on the Hamilton Rating Scale for Depression
* Able to tolerate psychotropic washout and no psychotropic medication, other than lorazepam (up to 3 mg/d PRN), during the study
* Recommended to receive ECT

Exclusion Criteria:

* History of schizophrenia, schizoaffective disorder, other functional psychosis, or rapid cycling bipolar disorder
* Secondary diagnosis of a delirium, dementia, or amnestic disorder, or epilepsy
* Pregnant
* History of neurological illness other than conditions associated with psychotropic exposure (e.g., tardive dyskinesia)
* History of alcohol or substance abuse within the year prior to study entry
* History of ECT within the 6 months prior to study entry

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 1998-12; Primary Completion 2002-12 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Short-term antidepressant efficacy | Measured immediately post-treatment and 2, 4, and 6 months post-treatment
  Primary outcome reflected change in HRSD depression symptom scores.
Specific acute, short-term, and long-term objective and subjective cognitive outcome measures (e.g., autobiographical amnesia, global self-rating of amnesia) | Measured immediately post-treatment and 2, 4, and 6 months post-treatment
  Specific neuropsychological measures were preselected as primary in safety analyses

SECONDARY OUTCOMES:
Antidepressant efficacy | Measured immediately post-treatment and 2, 4, and 6 months post-treatment
  Treatment groups were also compared in rates of response and remission, as well as post-treatment relapse.
Assessments of functional outcomes | Measured immediately post-treatment and 2, 4, and 6 months post-treatment
  Repeated measurement using the SF-36
Memory, non-memory, and executive functions (acute, short-term, and long-term measures) | Measured immediately post-treatment and 2, 4, and 6 months post-treatment
  Remaining measures in the neuropsychological battery other than those pre-selected as primary outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Harold A. Sackeim, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Result] Sackeim, H. A.: The convulsant and anticonvulsant properties of electroconvulsive therapy: towards a focal form of brain stimulation. Clinical Neuroscience Review, 2004, 4:39-57.
- [Result] Sackeim HA, Prudic J, Nobler MS, Fitzsimons L, Lisanby SH, Payne N, Berman RM, Brakemeier EL, Perera T, Devanand DP. Effects of pulse width and electrode placement on the efficacy and cognitive effects of electroconvulsive therapy. Brain Stimul. 2008 Apr;1(2):71-83. doi: 10.1016/j.brs.2008.03.001. PMID 19756236